CLINICAL TRIAL: NCT00896753
Title: Gene Expression Profiling of Metastatic Colon Cancer (CCCWFU 89B03)
Brief Title: Gene Expression Profiling in Normal Tissue and Tumor Tissue From Patients With Colon Cancer That Has Spread to the Liver, Lungs, or Peritoneum
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000550060; CCCWFU-89B03; CCCWFU-BG03-403
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2015-09

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage IV colon cancer; liver metastases; lung metastases; recurrent colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with metastatic colon cancer

SUMMARY:
RATIONALE: Studying the genes expressed in samples of tissue from patients with cancer may help doctors identify biomarkers related to cancer.

PURPOSE: This laboratory study is using gene expression profiling to evaluate normal tissue and tumor tissue from patients with colon cancer that has spread to the liver, lungs, or peritoneum.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate gene expression profiles in normal and tumor tissue from patients with colon cancer metastatic to the liver, lungs, or peritoneum.
* Establish cell lines from primary colon tumors metastatic to the liver, lungs, or peritoneum.
* Determine the specific gene expression changes that result in the manifestation of the drug-resistant phenotype for each metastatic site.

OUTLINE: This is a pilot study.

Tumor and normal tissue collected during surgery are analyzed for gene expression profiling by cDNA microarray. Tissue is also analyzed for thymidylate synthase (TS) gene expression by quantitative PCR and for protein expression by western blot. Gene expression patterns are correlated with TS levels.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of colon cancer metastatic to the liver, lungs, or peritoneum

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with metastatic colen cancer
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2003-09; Primary Completion 2006-09 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Gene expression changes that occur at each metastatic site (i.e., liver, lungs, and peritoneum) | day 1
Development of cell lines from primary colon tumors metastatic to the liver, lungs, or peritoneum | day 1

CONTACTS AND LOCATIONS:
Overall Officials: Perry Shen, MD, Study Chair — Wake Forest University Health Sciences